CLINICAL TRIAL: NCT03485989
Title: Role of Hazelnut Consumption in Improving Micronutrient Status in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon State University (Other)
Collaborators: Hazelnut Marketing Board (Unknown)
Responsible Party: Principal Investigator, Maret Traber, Professor, Oregon State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 6988
Record Dates: First submitted 2018-03-13; First posted 2018-04-03 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Nutrition Poor; Micronutrient Deficiency; Aging
Keywords: hazelnuts; vitamin E; aging
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hazelnuts (Experimental): Participants given 2 ounces (~57 grams) of dry roasted hazelnuts to consume each day.
  Interventions: Other: Hazelnuts

INTERVENTIONS:
Other: Hazelnuts — Dry roasted, individually packaged hazelnuts provided from the Hazelnuts Marketing Board of Oregon

SUMMARY:
With advancing age, older adults are susceptible to vitamin and mineral deficiencies for a variety of reasons. Nutrient-dense food sources of vitamin E and other key vitamins and minerals, like hazelnuts, may offer a simple means of improving nutritional status of healthy older adults.

This hypothesis is that individuals eating hazelnuts everyday will result in measurable increases in magnesium and vitamin E levels, two under-consumed micronutrients among older adults. Thus, subjects will consume two ounces (56 g) of hazelnuts each day for sixteen weeks. Investigators will measure vitamin E and magnesium levels along with a general assessment of micronutrient status as primary outcomes. Since nuts are nutrient-rich sources of unsaturated fatty acids but low in carbohydrates, changes in fasting glucose, lipid and lipoprotein profiles, and BMI will also be determined (secondary outcomes).

DETAILED DESCRIPTION:
Older adults are at increased risk of various chronic diseases where inadequate levels of vitamins and minerals may play a significant role, including cardiovascular disease, Alzheimer's disease, liver disease, and cancer. Older adults are increasingly more susceptible to vitamin and mineral deficiencies with changes in dietary preferences, changes in socioeconomic status, decreased consumption of a variety of foods, poor absorption in the gut, and an increased demand for many of these micronutrients with advanced age.

Epidemiological studies and recent clinical trials have shown that use of multivitamin/mineral or single nutrient supplements, such as vitamin E, have beneficial effects on disease risk, but many people are hesitant to use dietary supplements due to reports of ineffectiveness or potential negative effects. However, food sources of vitamin E and other key vitamins and minerals continue to show health benefits. As an alternative to mandating consumption of multivitamin and mineral supplements or food fortification, a dietary solution is to increase consumption of nutrient-dense foods, like hazelnuts.

Tree nuts, including hazelnuts, contain a wide variety of vitamins and minerals, and are particularly good source of vitamin E and magnesium, two "shortfall nutrients" that are lacking in the typical American diet. Over 90% of U.S. adults do not meet recommended intake levels of vitamin E, and 60% do not get enough magnesium. Tree nuts are also a good source of protein and fiber and are high in healthful unsaturated fatty acids and phytochemicals such as flavonoids and phytosterols.

Most clinical studies on the benefits of nut consumption have been conducted using almonds and walnuts, with hazelnuts used less frequently. However, the health benefits of consuming hazelnuts have been demonstrated in many clinical trials, including lower blood glucose levels, alterations in blood lipids, and declines in biomarkers of oxidative stress. Although several clinical trials have investigated nutritional impact of hazelnuts in adults, no clinical trials with hazelnuts have focused on examining micronutrient status and potential health benefits only in older (≥55 years) adults.

Determination of body status of many micronutrients can be difficult, especially so the evaluation of vitamin E levels when age is considered as a factor. Although serum α-tocopherol levels are generally higher in adults above the age of 50 compared to younger adults, the increased prevalence of hypercholesterolemia in older adults makes interpretation of circulating α-tocopherol levels difficult. Alternatively, urinary α- and γ-carboxyethyl hydroxychromanol (α- and γ-CEHC) is believed to be a biomarker of α- and γ-tocopherol status that changes with vitamin E intake. In particular, low α-CEHC excretion is considered a reliable marker of poor α-tocopherol status, while an increase in α-CEHC is indicative of adequate α-tocopherol status.

The objective of this study was to determine whether daily hazelnut consumption by healthy older adults for 16 weeks improves biomarkers of micronutrient status, especially vitamin E and magnesium. For a detailed assessment of vitamin E status, plasma α- and γ-tocopherol concentrations were determined together with urinary α- and γ-CEHC levels. In addition, a commercially available lymphocyte proliferation assay was utilized to evaluate the status of several other micronutrients. Since hazelnut consumption is reported to reduce blood lipids and improve glucose homeostasis, these biomarkers were also monitored in our study.

ELIGIBILITY:
Inclusion Criteria:

* Must be generally healthy
* Women must be post-menopausal (12 months period-free) or surgically sterile.
* Must be willing to eat two ounces (56 g) of dry roasted hazelnuts each day during the study
* Must refrain from taking nutritional supplements during the study
* Must follow a diet that excludes all nuts (other than those supplied), seeds, and other vitamin E-rich foods (see Restricted Foods and Supplements document)
* Must be willing to complete food frequency questionnaires
* Must be willing to give blood samples on 3 separate occasions and urine on 2 separate occasions

Exclusion Criteria:

* Current or past (two years) use of any tobacco (including e-cigarettes) and marijuana products
* Allergy to any nut including tree nuts and peanuts, or hazelnut pollen
* History of asthma
* Vitamin E supplement use during the last three months or regular use of vitamin E-enriched nutritional drinks (e.g. Ensure)
* Regular nut eaters: individuals that regularly consume > 3.5 ounces (112 g) of almonds, hazelnuts and/or sunflower seeds per week in any form (e.g. nuts, nut butters, nut oil, etc.), and no more than 10 mg alpha-tocopherol (vitamin E) per day from their diet.
* Bariatric surgery (e.g. gastric bypass, gastric banding, sleeve gastrectomy, etc.), or serious chronic illness including Crohn's disease, celiac disease, diverticulitis, chronic diarrhea, ulcerative colitis, gastritis
* History of cardiovascular disease including stroke, heart attack, or congestive heart failure
* Any history of arterial bypass or stent placement.
* History of emphysema or chronic obstructive pulmonary disease (COPD)
* Stage II hypertension (either systolic pressure > 159 mm Hg or diastolic pressure 99 mm Hg)
* History of cancer during the previous 5 years
* Diabetes (type 1 or type 2) or use of drugs to lower blood sugar or increase insulin production or sensitivity
* Use of medications to lower cholesterol other than statins
* Use of medications to decrease fat or cholesterol absorption
* Unwillingness to refrain from taking dietary supplements (except calcium and vitamin D and vitamin B12), magnesium-containing drugs such as certain antacids, stool softeners and laxatives
* BMI < 18.5 or > 35
* Blood chemistry limits; any of the following at screening excludes participation:

  * Fasting blood glucose ≥ 126 mg/dL
  * LDL cholesterol ≥160 mg/dL
  * Triglyceride ≥200 mg/dL
  * High-sensitivity C-reactive protein (hsCRP) > 10 mg/L

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2017-12-29 (Actual)

PRIMARY OUTCOMES:
Changes in Plasma Micronutrient Levels | Between baseline (Visit 2) and 16 weeks (last visit)
  Plasma levels of magnesium and vitamin E (alpha and gamma tocopherol) at baseline and 16 weeks after hazelnut intervention will be determined. Vitamin E analyses will be performed as absolute concentrations and concentrations corrected for total plasma lipids.
Changes in Plasma Urine Vitamin E Metabolites | Between baseline (Visit 2) and 16 weeks (last visit)
  Urine concentrations of alpha and gamma carboxyethyl hydroxychroman (metabolites of alpha and gamma tocopherol, respectively) will be determined at baseline and 16 weeks after hazelnut intervention. Urine values will be corrected for creatinine levels.
Changes in Lymphocyte Proliferation Assay | Between baseline (Visit 2) and 16 weeks (last visit)
  Blood samples will be collected and sent to Spectracell Labs, Inc. for a functional micronutrient analysis utilizing their proprietary lymphocyte proliferation assay. Micronutrient levels in these white blood cell samples will be assessed by changes in lymphocyte proliferation in the absence of a given vitamin or mineral, suggesting functional inadequacies that may not correspond to plasma values. Data will be represented as percent difference in cell proliferative capacity in cells growing in a complete media vs. a single-nutrient deprived media.

SECONDARY OUTCOMES:
Lipid Status | Between baseline (Visit 2) and 16 weeks (last visit)
  Lipid profile will be determined from samples blood sent to a CLIA(Clinical Laboratory Improvement Amendments)-certified laboratory. Changes to fasting lipoprotein and triglyceride status determined before and after hazelnut intervention.
Glucose Homeostasis | Between baseline (Visit 2) and 16 weeks (last visit)
  Glucose and insulin levels will be determined from blood samples to a CLIA-certified laboratory. Changes to fasting glucose levels and insulin levels determined before and after hazelnut intervention.
BMI | Between baseline (Visit 2) and 16 weeks (last visit)
  Height and weight will be measured by stadiometer and scale. Changes to height and weight will be expressed as BMI calculated before and after hazelnut intervention.
Blood Pressure | Between baseline (Visit 2) and 16 weeks (last visit)
  Changes to resting systolic and diastolic blood pressure (mmHg) will be measured by sphygmomanometer before and after hazelnut intervention.
Heart Rate | Between baseline (Visit 2) and 16 weeks (last visit)
  Resting heart rate will be measured manually using the ventral aspect of radial artery.

CONTACTS AND LOCATIONS:
Overall Officials: Maret G Traber, PhD, Principal Investigator — Oregon State University
Locations (1):
- Linus Pauling Science Center, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Michels AJ, Leonard SW, Uesugi SL, Bobe G, Frei B, Traber MG. Daily Consumption of Oregon Hazelnuts Affects alpha-Tocopherol Status in Healthy Older Adults: A Pre-Post Intervention Study. J Nutr. 2018 Dec 1;148(12):1924-1930. doi: 10.1093/jn/nxy210. PMID 30517727